CLINICAL TRIAL: NCT02746614
Title: Psychomotor Therapy Effects Adaptive Behavior and Motor Proficiency of Adults With Intellectual Disability
Brief Title: Psychomotor Therapy Effects in Adaptive Behavior and Motor Proficiency in Intellectual Disability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Faculdade de Motricidade Humana (Other)
Responsible Party: Principal Investigator, Sofia Santos, PhD, Faculdade de Motricidade Humana
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: FaculdadeMH
Record Dates: First submitted 2016-04-04; First posted 2016-04-21 (Estimated); Last update posted 2016-04-21 (Estimated); Status verified 2016-04

CONDITIONS: Intellectual Disability
Keywords: adaptive behavior; motor proficiency; psychomotor therapy; intellectual disability
MeSH Terms: conditions — Intellectual Disability

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Psychomotor Therapy & Adaptive Behavior (Active Comparator): After the initial assessment of adaptive behavior, i.e.., set of skills that each individual with intellectual disability should train to cope with environmental demands, a Psychomotor Intervention Program was designed specifically. The program integrated individual and group sessions during 3 months, and the main goals of the program were related to independent functioning, motor development, economic and professional activities, academic and verbal skills.
  Interventions: Other: Psychomotor Therapy
- Psychomotor Therapy & Motor Proficiency (Active Comparator): Motor Proficiency After the initial assessment, a Psychomotor Intervention Program was designed specifically for participants with IDD. This program integrated individual and group sessions during 3 months, and the main goals of the program were related to motor coordination (balance, manual dexterity and coordination, global and fine praxis).
  Interventions: Other: Psychomotor Therapy

INTERVENTIONS:
Other: Psychomotor Therapy — Psychomotor Therapy

SUMMARY:
People with intellectual and developmental disabilities (IDD) usually present limitations at adaptive behavior and motor skills, which lead to limitations/barriers in the daily independent functioning of this population. The main goal of this research is to analyze the efficacy of a Psychomotor Intervention Program on adults with and without IDD, through an assessment of their progress both in adaptive behavior competences and motor proficiency skills.

DETAILED DESCRIPTION:
This study sample comprised 15 participants divided by three groups of 5 individuals each: one group with IDD (with different ethiology), another one with Down Syndrome and the third with typical development. Ages range from 22 to 31 years-old (Average=26,5; St. Deviation=3,76), 6 were females and 9 males. All adults with IDD were all institutionalized at an Occupation Activities Centre of an institution and adults without ID were selected by convenience, with ages comprised within the selected range. All groups were compared through both evaluation instruments: the Portuguese version of Adaptive Behavior Scale (PABS) and Bruininks-Oseretsky Motor Proficiency Test (BOT-2). Both tests were applied according to original protocols. Ethics requisites were fulfilled. After the initial assessment, a Psychomotor Intervention Program was designed specifically for participants with IDD. This program integrated individual and group sessions during 3 months, and the main goals of the program were related to motor coordination (balance, manual dexterity and coordination, global and fine praxis), economic and professional activities, academic and verbal skills.

ELIGIBILITY:
Inclusion Criteria:

* ages above 18 years
* diagnosis of intellectual disability
* institution in Castelo Branco

Exclusion Criteria:

* other co-morbilities associated
* not institutionalised

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2014-09; Primary Completion 2015-07 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Test of Motor Proficiency of Bruininski-Oseretsky 2 | one year
Portuguese Adaptive Behavior Scale | one year

IPD SHARING:
Plan to Share IPD: Yes
All individual data were provided to institutions where the individuals were, helping in Individual Program' planning